CLINICAL TRIAL: NCT04498026
Title: A Pivotal Clinical Trial Evaluating the Safety and Effectiveness of Adherus™ AutoSpray and Adherus™ AutoSpray ET Dural Sealant When Used as a Dural Sealant in Spinal Procedures
Brief Title: Adherus™ Dural Sealant in Spinal Procedures
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Craniomaxillofacial (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HBMT-US-2019-001
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Spinal Duraplasty
Keywords: Adherus Dural Sealant; Adherus AutoSpray Dural Sealant; Dura mater; Durotomy; CSF leak
MeSH Terms: conditions — Cerebrospinal Fluid Otorrhea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Adherus Dural Sealant System (Experimental): Device: Adherus Dural Sealant, In situ polymerizing sealant
  Interventions: Device: Adherus Dural Sealant System
- DuraSeal Exact Dural Sealant System (Active Comparator): Device: DuraSeal Exact (P080013b)
  Interventions: Device: DuraSeal Exact Dural Sealant System

INTERVENTIONS:
Device: Adherus Dural Sealant System — Adherus Dural Sealant, In situ polymerizing sealant
  Arms: Adherus Dural Sealant System
Device: DuraSeal Exact Dural Sealant System — DuraSeal Exact (P080013b)
  Arms: DuraSeal Exact Dural Sealant System

SUMMARY:
The purpose of this study is to test an experimental device, the Adherus AutoSpray and Adherus AutoSpray ET Dural Sealant, in spinal surgical procedures.

This study is being done to compare Adherus AutoSpray and Adherus AutoSpray ET Dural Sealant to DuraSeal Exact Spinal Sealant, which has already received Federal Food and Drug Administration (FDA) approval in spinal procedures.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, single-blind, multicenter, pivotal trial that will evaluate the safety and effectiveness of Adherus Dural Sealant when used in conjunction with standard methods of dural repair in spinal procedures. This trial uses the commercially available DuraSeal Exact as an active control. The trial is designed to demonstrate non-inferiority of Adherus Dural Sealant to DuraSeal Exact.

Subjects who are undergoing spinal surgery, consent to participate in this trial and experience a durotomy will be considered for study enrollment. Following a two-tiered inclusion/exclusion consideration, subjects will be randomized intraoperatively using a 1:1 randomization ratio. Up to 90 subjects will be randomized to treatment with either Adherus Dural Sealant or DuraSeal Exact with at least 50% of subjects undergoing procedures at lumbar or lumbosacral levels. Up to 30 investigational sites within the United States will participate in this trial.

A primary composite endpoint evaluating safety and effectiveness will be measured within a 90-day required follow-up period post-procedure. Subjects will be followed at discharge or between postoperative days (POD) 1-4 from the index procedure (whichever occurs first) and at 30 days and 90 days post-index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 and ≤ 75 years old.
2. Subject is scheduled for an elective spinal procedure that will require a planned durotomy.
3. Subject requires a procedure involving a Class I/clean wound (uninfected surgical wound in which no inflammation is encountered).
4. Subject is able and willing to provide informed consent and HIPAA authorization.
5. Subject is able and willing to meet all study requirements, including attending all post-index procedure assessment visits and radiological tests.

   Intra-Operative Inclusion Criteria:
6. Subject has durotomy edges that can be re-approximated using the investigator's standard methods of dural repair.

Exclusion Criteria:

1. Subject has clinically significant hydrocephalus or clinical evidence of altered CSF dynamics.
2. Subject has a pre-existing external lumbar CSF drain or internal CSF shunt.
3. Subject has experienced previous CSF leak (secondary to trauma, neoplasm, surgery, or other etiology).
4. Subject is undergoing a Chiari malformation procedure.
5. Subject has undergone a previous spinal procedure in the same anatomical location.
6. Subject has had radiation treatment to the surgical site, or standard fractionated radiation therapy is planned within ten days post indexprocedure.
7. Subject has spinal metallic implants that may cause significant imaging artifact on the MRI evaluation of the spine.
8. Subject has metallic implant(s) that are not MRI compatible, e.g., cochlear implant, neurostimulator, stent, surgical clip, cardiac pacemakers, or other non-MRI compatible implants, or an elective implant of such devices is planned during the course of the study. Note: mercury amalgam dental fillings or similar metallic dental prostheses are not an exclusion criterion.
9. Subject has a known malignancy or another condition with anticipated survival shorter than six months.
10. Subject has undergone chemotherapy treatment, excluding hormonal therapy, within three weeks prior to the planned index procedure, or chemotherapy treatment is planned within two weeks after the index procedure is performed.
11. Subject has been treated with chronic steroid therapy (defined as regular (daily) administration of steroid agent(s) for ≥ 8 weeks) unless discontinued greater than four weeks prior to the planned index procedure. Note: standard acute perioperative steroids are permitted; administration of steroid agents for < 8 weeks duration prior to the planned index procedure is permitted.
12. Subject has received warfarin, heparin, other anticoagulant agents, aspirin or non steroid anti-inflammatory agents on a daily basis and pre-surgical, standard of care drug wash-out did not occur.
13. Subject has a compromised immune system or autoimmune disease or is on chronic immunosuppressant agents at baseline.
14. Subject has a systemic infection or evidence of any infection near planned operative site.
15. Subject has a serum creatinine level > 2.0 mg/dL.
16. Subject has a serum total bilirubin > 2.5 mg/dL at baseline.
17. Subject has uncontrolled diabetes as evidenced by an HbA1c > 7% prior to surgery.
18. Subject has a known allergy to FD&C Blue #1 and/or FD&C Yellow #5 or any of the constituents of the dural sealants.
19. Subject is pregnant, breast-feeding, or intends to become pregnant during the course of the study.
20. Subject is participating in a clinical trial of another investigational drug or device and has not completed the required follow-up period.

    Intra-Operative Exclusion Criteria:
21. Subject has an incidental finding that meets any pre-operative exclusion criterion listed above.
22. Subject's dural defect cannot be closed with suture and/or duraplasty material.
23. Subject has a gap > 2 mm present between dural edges, or between the edge of dura and duraplasty material, based on visual estimate by surgeon before application of the surgical sealant.
24. Subject had undergone laminoplasty decompression.
25. Subject had undergone a syringomyelia procedure where the shunt is not placed in the subarachnoid position.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of treated subjects who are free from the following incidences: | 90 Days
  * CSF leak or pseudomeningocele diagnosed by physical examination, biochemical assay or imaging study during the 90-day follow-up period following the index procedure
  * Unplanned retreatment of the original surgical site adjudicated by the Clinical Events Committee (CEC) to be device-related, other than CSF leak or pseudomeningocele formation or those related to the subject's pre-existing condition, during the 90-day follow-up period including:
    * treatment for deep infection
    * treatment for meningitis
    * minimally invasive procedures or return to the operating room for neurosurgical complications

SECONDARY OUTCOMES:
Secondary endpoints, which will only be tested for superiority of Adherus over DuraSeal Exact after the primary objective of the study has been met: | 30 Day, 90 Day
  * CSF leak or pseudomeningocele diagnosed by physical examination, biochemical assay or imaging study during the 30-day and 90-day follow-up period following the index procedure
  * Unplanned retreatment of the original surgical site adjudicated by the CEC to be device-related, other than CSF leak or pseudomeningocele formation or those related to the subject's pre-existing condition, during the 30-day and 90-day follow-up period including:
    * treatment for deep infection
    * treatment for meningitis
    * minimally invasive procedures or return to the operating room for neurosurgical complications

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - City of Hope National Medical Center, Duarte, California
  - University of California Davis Health, Sacramento, California
  - Stanford University, Stanford, California
  - Mayo Clinic (FL), Jacksonville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Irving Medical Center, New York, New York
  - Carolina Neurosurgery & Spine Associates, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Houston Methodist Research Institute, Houston, Texas
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Carilion Clinic, Roanoke, Virginia